CLINICAL TRIAL: NCT00201149
Title: Hypertension Control and Therapy Adherence
Brief Title: Clinician Counseling and Cultural Competency to Improve Hypertension Control and Therapy Adherence
Acronym: HCTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nancy Kressin, BMC Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 255; R01HL072814 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): In one team of clinicians we will implement only the patient-centered counseling program.
  Interventions: Behavioral: Patient-centered Counseling
- 3 (No Intervention): The control group will provide usual care
- 2 (Experimental): In a subset of those clinicians receiving the patient-centered counseling program intervention, we will augment it with cultural competency training.
  Interventions: Behavioral: Patient-centered Counseling

INTERVENTIONS:
Behavioral: Patient-centered Counseling — To improve patients' adherence with prescribed anti-hypertensive medication, improve blood pressure control and doctor-patient communication, we propose a three-armed randomized controlled trial in the internal medicine clinics of a large metropolitan teaching hospital which serves a large percentage of poor African American and white patients. We will implement an intervention strategy by teaching clinicians to counsel patients about hypertension control through the use of patient-centered counseling and by providing office-based support; critical to facilitating clinicians' use of this strategy. Through this intervention we will provide clinicians with communication skills that are proven to help patients change risk-related behaviors, and which will enhance doctor-patient communication.
  Arms: 1; 2

SUMMARY:
The purpose of this study is to test the effect of clinician counseling and cultural competence training on medication compliance and blood pressure (BP) control in patients with high BP.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension affects nearly 50 million people in the U.S. and is related to increased medical morbidity and mortality associated with a range of medical disorders. Despite the availability of effective treatments for BP control, less than 25 percent of patients with hypertension demonstrate such control, and researchers have found this to be related to important patient factors associated with pharmacotherapy adherence. Further, research has demonstrated that this adherence problem is greater among African Americans than among Caucasians. The focus of the study is on improvements in adherence among patients with hypertension. The study is most specifically targeted to reducing racial disparities in medication adherence by including an interventional element that specifically targets African American patients in its approach.

DESIGN NARRATIVE:

To improve patients' adherence with prescribed anti-hypertensive medication, BP control, and doctor-patient communication, and to decrease racial disparities in each area, the investigators will conduct a three-armed randomized controlled study in the general internal medicine clinics of a large urban teaching hospital serving many poor African American and white patients. Proven intervention strategies will be implemented by teaching clinicians to use patient-centered counseling, enhancing skills that are known to help patients change health-related behaviors, and enhancing cultural competency among clinicians, thereby further improving clinician-patient communication. One group of clinicians will implement only the patient-centered counseling program. A second group will implement the patient-centered counseling education program, augmenting it with an established method for cultural competency training. A third group (control group) will provide usual care. To assess outcomes, the study will evaluate pre-intervention patient adherence to prescribed medications through patient self-report and the use of electronic pill top monitoring, clinicians' provision of advice and counseling about anti-hypertensive medications and use of cultural competency skills, and the proportion of patients with controlled BP. Subsequent to the interventions, each of these outcomes will be assessed.

The aims of this study are to: 1) improve patients' adherence to prescribed anti-hypertensive therapy; 1a. examine adherence rates at baseline, and examine whether there are racial differences in adherence; 1b. decrease racial disparities in patient adherence with anti-hypertensive therapy from the baseline to the follow-up assessments; and 1c. evaluate the relative efficacy of the patient-centered counseling intervention compared to patient-centered counseling augmented by cultural competency training on patients' medication adherence; 2) increase the proportion of patients with controlled hypertension; 2a. examine the baseline proportion of patients with controlled hypertension, and whether there are racial differences in rates of control; 2b. decrease racial disparities in the proportion of patients with controlled hypertension from the baseline to the follow-up assessments; and 2c. evaluate the relative efficacy of patient-centered counseling compared to patient-centered counseling augmented by cultural competency training on patients' BP control; and 3) improve clinicians' communication with patients regarding medication use, as measured by increased frequency of clinicians' provision of advice and counseling about anti-hypertensive medications and use of culturally competent communication styles; 3a. examine whether there are racial disparities in clinicians' provision of advice and counseling or culturally competent communication patterns about anti-hypertensive medications at baseline; 3b. examine whether the proposed interventions decrease any observed racial disparities in clinician communication over time; and 3c. evaluate the relative efficacy of the patient-centered counseling intervention compared to patient-centered counseling augmented by cultural competency training on clinicians' communication patterns.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for care at least once in the General Internal Medicine clinic
* Diagnosis of hypertension, as listed on a medical problem list or elsewhere within the medical record
* Already prescribed antihypertensive medications

Exclusion Criteria:

* Musculoskeletal problems preventing successful opening of the electronic pill tops
* Cognitive status limitations, including psychiatric disorders such as schizophrenia
* Active alcohol or substance abuse problems
* Does not speak English

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2004-02; Primary Completion 2008-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient medication adherence (self-reported at baseline and follow-up visit [6-9 months after initial recruitment]and measured with electronic monitoring caps 90 days after baseline visit and 90 days after follow-up visit) | September 2004 - May 2008
Proportion of patients with controlled hypertension (measured at baseline and follow-up visit [6-9 months after initial recruitment]) | September 2004 - May 2008
Use of communication strategies by clinicians (measured at baseline and follow-up visit [6-9 months after initial recruitment]) | September 2004 - May 2008

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nancy Kressin, Study Chair — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manze MG, Orner MB, Glickman M, Pbert L, Berlowitz D, Kressin NR. Brief provider communication skills training fails to impact patient hypertension outcomes. Patient Educ Couns. 2015 Feb;98(2):191-8. doi: 10.1016/j.pec.2014.10.014. Epub 2014 Oct 27. PMID 25468397
- See also: 1. Rose, A, Glickman, ME, D'Amore, MM, Orner, MB, Berlowitz, D, Kressin, NR. (2011). Effects of Daily Adherence to Anti-Hypertensive Medication on Blood Pressure Control. Journal of Clinical Hypertension: Jun; 13(6): 416-21 — http://onlinelibrary.wiley.com/doi/10.1111/j.1751-7176.2011.00427.x/full
- See also: 2. Kressin, NR, Orner, MB, Manze, M, Glickman, ME, Berlowitz, D. (2010). Understanding contributors to racial disparities in blood pressure control. Circulation: Quality and Outcomes: Mar;3(2):173-80. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2841788/?tool=pubmed
- See also: 3. Manze, M, Rose, AJ, Orner, MB, Berlowitz, DR, Kressin, NR (2010). Understanding Racial Disparities in Treatment Intensification for Hypertension Management. Journal of General Internal Medicine; 25 (8), 819-25. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2896595/?tool=pubmed
- See also: 4. Rose, AJ, Berlowitz, DR, Manze, M, Orner, MB, Kressin, NR (2009). Comparing methods of measuring treatment intensity in hypertension care. Circulation: Quality and Outcomes: 2; 385-391 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2801893/?tool=pubmed
- See also: 5. Rose, AJ, Berlowitz, DR, Manze, M, Orner, MB, Kressin, NR (2009). Intensifying Therapy for Hypertension Despite Suboptimal Adherence. Hypertension: 54(3): 524-529. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2739677/?tool=pubmed